CLINICAL TRIAL: NCT06324539
Title: Validation of a New Innovative Method for the Easy Detection of a Disease Specific Marker to Make Prompt Diagnosis of Celiac Disease in All the Clinical Manifestations: a Paediatric Multicenter Study.
Brief Title: Validation of a New Innovative Method for Specific Marker Detection in Celiac Disease
Status: Recruiting | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: PNRR-POC-2022-12376280
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Celiac Disease in Children
Keywords: Celiac disease; Intestinal antibodies; Rapid test
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood and biopsies samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Celiac Disease subjects
  Interventions: Diagnostic Test: Diagnostic Test: Rapid Intestinal anti-TG2 Assay
- Controls subjects
  Interventions: Diagnostic Test: Diagnostic Test: Rapid Intestinal anti-TG2 Assay

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: Rapid Intestinal anti-TG2 Assay — Evaluation of the reliability of the Rapid Intestinal anti-TG2 Assay for revealing anti-TG2 antibodies in duodenal biopsy specimens of patients suffering from CD, especially potential CD in which the diagnosis may be challenging.
  Intestinal anti-TG2 will be investigated also in patients suffering from other non-CD related gastrointestinal disorders. Sensitivity, specificity and likelihood ratios of the Rapid Intestinal anti-TG2 assay will be calculated and compared to the reference standard (serology + histopathology) of CD diagnosis.
  Groups: Celiac Disease subjects
Diagnostic Test: Diagnostic Test: Rapid Intestinal anti-TG2 Assay — Evaluation of the reliability of the Rapid Intestinal anti-TG2 Assay for revealing anti-TG2 antibodies in duodenal biopsy specimens of patients suffering from CD, especially potential CD in which the diagnosis may be challenging.
  Intestinal anti-TG2 will be investigated also in patients suffering from other non-CD related gastrointestinal disorders. Sensitivity, specificity and likelihood ratios of the Rapid Intestinal anti-TG2 assay will be calculated and compared to the reference standard (serology + histopathology) of CD diagnosis.
  Groups: Controls subjects

SUMMARY:
Celiac disease (CD) is a common auto-immune disorder induced by gluten ingestion in genetically susceptible individuals (HLA-DQ2/DQ8). Gluten induces small-bowel villous atrophy and a specific immune response characterized by the production of CD-autoantibodies against transglutaminase 2 (anti-TG2) and endomysium (EMA). In symptomatic patients with positive-serum antibodies and villous atrophy, the diagnosis of CD is clearcut.

However, 10-30% of patients evaluated for suspected CD show only mild histopathologic changes and fluctuating serologic markers, a condition identified as potential CD. In such cases the diagnosis may remain uncertain.

CD-autoantibodies are produced by intestinal B-cells in the early phases of the disease, before their appearance in the serum and when the duodenal mucosa is still normal. Intestinal CD-antibodies (I-CD-abs) are a marker of CD, have a high sensitivity and specificity for CD and identify those patients with potential CD who are at risk of progression to villous atrophy. I-CD-abs can be detected by double immunofluorescence staining on frozen duodenal sections or by using an endomysial antibody assay in the culture medium of duodenal biopsies (EMAbiopsy).

The diagnostic accuracy of these techniques is comparable as they both have high sensitivity and specificity. However, their implementation in clinical practice is limited because they require both experienced operators and well-equipped laboratories. There is an unmet need: the development of a new simple and effective diagnostic tool that any gastroenterology unit can use in routine diagnostics to ensure a prompt diagnosis in suspected CD patients, who may benefit from a therapy based on gluten-free diet, and to reduce both unnecessary medical investigations and diagnostic delays.

In order to simplify and shorten times for the detection of these intestinal antibodies, the study aims to substitute the EMAbiopsy assay with a supernatant obtained quickly after mechanical lysis of fresh intestinal biopsy specimen. The obtained samples will be tested with rapid (about 15 minutes) immune-chromatographic anti-TG2 assay (Rapid Intestinal anti-TG2 Assay).

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing an elective esophagogastroduodenoscopy (EGD) for suspected Celiac Disease (CD), eosinophilic esophagitis, autoimmune enteropathy, inflammatory bowel disease, gastritis, gastric or duodenal ulcer, gastroesophageal reflux disease.

Exclusion Criteria:

* Bleeding disorders
* Patients fulfilling the new European Society for Paediatric Gastroenterology Hepatology and Nutrition (ESPGHAN) guidelines for diagnosing CD (version 2020) for a serology-based CD diagnosis
* Subjects in whom intestinal biopsies are not indicated as part of the diagnostic process

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children (aged between 2 and 17 years) referred to the Gastroenterology Units for elective gastro-intestinal endoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 332 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the EMA-biopsy in comparison to the reference standard (serology + histology) for CD diagnosis | Through study completion, an average of 18 months
Specificity of the EMA-biopsy in comparison to the reference standard (serology + histology) for CD diagnosis | Through study completion, an average of 18 months
Sensitivity of the Rapid Intestinal anti-TG2 Assay in comparison to the reference standard (serology + histology) for CD diagnosis | Through study completion, an average of 18 months
Specificity of the Rapid Intestinal anti-TG2 Assay in comparison to the reference standard (serology + histology) for CD diagnosis | Through study completion, an average of 18 months

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Consorzio per Valutazioni Biologiche e Faramacologiche, Pavia
  - Azienda ULSS2 Marca Trevigiana, Treviso
  - Institute for Maternal and Child Health - IRCCS "Burlo Garofolo", Trieste

IPD SHARING:
Plan to Share IPD: Undecided